CLINICAL TRIAL: NCT01962844
Title: The Effect of Extra Virgin Coconut Oil Treatment Nutritional Associated With Data Anthropometric and Lipid Profile in Patients With Chronic Heart Disease
Brief Title: Coconut Oil in Cardiovascular Disease
Acronym: HCCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, DIULI ALVES CARDOSO, researcher official, Universidade Federal do Rio de Janeiro
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FC 0305
Record Dates: First submitted 2013-10-08; First posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Coronary Artery Disease
Keywords: chronic coronary artery disease; coconut oil extra virgin; index of diet quality; nutritional treatment
MeSH Terms: interventions — Coconut Oil; Diet; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutritional treatment (Other): All patients received an individualized diet plan and balanced. The diet was calculated according to the nutritional status and the protein 15-20% of total energy value, lipids 25-30% of daily energy intake and carbohydrate 50-60% of of total energy value
  Interventions: Behavioral: Diet
- extra virgim coconut oil group (Experimental): Oil from coconuts (cocos nucifera L.) contains a high proportion of medium chain fatty acids, principally the lauric acid (12:0), in proportions that range from 45 to 50%
  Interventions: Dietary Supplement: Coconut Oil

INTERVENTIONS:
Dietary Supplement: Coconut Oil — Patients were followed for 6 months with dietary treatment. Beginning supplementation with coconut oil extra virgin from the third month of intervention nutrition. Coconut oil was consumed neat or added to fruit.
  Other Names: coconut oil, palm grease, palmoil
  Arms: extra virgim coconut oil group
Behavioral: Diet — Patients were instructed to follow the dietary treatment for 6 months
  Other Names: dietary advice
  Arms: Nutritional treatment

SUMMARY:
The purpose of this study is to evaluate the supplementation with extra virgin of coconut oil combined with a nutritional counseling in reducing anthropometry and improves the lipid profile in patients with chronic coronary disease.

DETAILED DESCRIPTION:
The universe of patients with coronary artery disease (CAD) has been increasing steadily worldwide. And associated intimately with certain cardiovascular risk factors such as dyslipidemia , decreased HDL-C , hypertension , diabetes mellitus and obesity. The quality of the fat in the diet influences the incidence of obesity and dyslipidemia. A high intake of saturated fat in different populations is associated with elevated serum cholesterol concentration and cardiovascular mortality. However, studies have shown that extra virgin coconut oil (Cocos nucifera L.) despite being characterized by its high content of saturated fat was not associated with obesity and dyslipidemia in populations that had their high consumption . And this is due to the high proportion of medium chain triglycerides , especially lauric acid in proportions ranging from 45-50 % , and the presence of factors antioxidants like vitamin E and polyphenols. Our hypothesis is that extra virgin coconut oil associated with a nutritional treatment has an effect on weight reduction and control of dyslipidemia contributes to control in secondary prevention in patients with coronary artery disease. All participants will be informed about the research and they must sign a consent form . Volunteers will be divided into two groups : a group receiving dietary treatment for 6 months and the other beyond the dietary treatment during the 6 months starts to receive supplementation with coconut oil extra virgin from 3 months, both groups evaluated monthly . At each visit , weight assessment , compliance with diet and blood pressure measurement is performed. In addition , the blood will also be collected for determination of glucose, insulin, total cholesterol, LDL-cholesterol , HDL-cholesterol, triglycerides , apolipoprotein A and B. The results will be analyzed by the statistical program.It is expected that the results obtained, the extra virgin coconut oil can be used as a coupled secondary prevention in patients with coronary artery disease.Our hypothesis is that extra virgin coconut oil associated with nutritional treatment has an effect on weight reduction and control of dyslipidemia contributes to control in secondary prevention in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

Presenting chronic coronary artery disease (myocardial infarction and/or stable angina

Exclusion Criteria:

angioplasty and/or coronary artery bypass grafting and previous cardiovascular event <6 months and those who had chronic renal failure with creatinine values> the 2mg/dl and liver disease.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Anthropometry | 3 months
  To evaluate the effect of extra virgin coconut oil in the improvement of weight, waist circumference and neck circumference in patients with chronic coronary artery disease

SECONDARY OUTCOMES:
Lipid profile | 3 months
  To evaluate the effect of extra virgin coconut oil in lowering total cholesterol, triglycerides, LDL cholesterol and increase in HDL cholesterol
Quality of the diet | 3 months
  To evaluating the effect of treatment on the nutritional quality of the diet

CONTACTS AND LOCATIONS:
Overall Officials: Diuli A Cardoso, Ms, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Instituto Nacional do Coração, Rio de Janeiro, Rio de Janeiro, Brazil